CLINICAL TRIAL: NCT06806982
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of VRN101099 in Patients With HER2-Positive Solid Tumors
Brief Title: A Study of VRN101099 in Patients With HER2-Positive Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Voronoi, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRN101099_01
Record Dates: First submitted 2025-01-06; First posted 2025-02-04 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: HER2-positive Solid Tumors
Keywords: HER2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VRN101099 (Experimental): VRN101099 capsules will be administered orally as monotherapy once daily over 21-day cycles Dose and frequency of dosing: The planned doses for dose escalation are 80 mg, 160 mg, 240 mg, 320 mg, 400 mg, and 480 mg once daily.
  Dosage form- Oral capsules
  Interventions: Drug: VRN101099

INTERVENTIONS:
Drug: VRN101099 — Oral capsules

SUMMARY:
This FIH open-label study aims to investigate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and antitumor effect of VRN101099 in patients with HER2-positive solid tumors for whom no standard therapies are available.

DETAILED DESCRIPTION:
This is an open-label study where eligible patients will receive VRN101099 capsules orally, once daily (QD) at the specified dose level, in repeated 21-day treatment cycles until disease progression (PD), death, loss to follow-up, start of another anticancer treatment, intolerable toxicity, withdrawal of consent, or study completion or closure (whichever occurs first).

Dose limiting toxicities (DLTs) will be monitored during the first cycle of treatment (i.e., 21 days of IP administration, Cycle 1).

The proposed VRN101099 dose levels are: 80 mg QD, 160 mg QD, 240 mg QD, 320 mg QD, 400 mg QD, and 480 mg QD.

Safety Monitoring committee will be setup for review DLTs and overall safety data. Border medical oncology in Australia will be using Omico for CaSP NGS screening participants to the study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years (patients in Korea must be aged ≥ 19 years).
2. Able to comprehend and willing to sign an informed consent form and to abide by the study requirements and restrictions.
3. Has at least 1 evaluable lesion (measurable or non-measurable) based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 (note: metastatic brain lesions will also be assessed using the Response Assessment in Neuro-Oncology - Brain Metastases [RANO-BM] as an exploratory objective).
4. Has confirmed HER2-positive or mutated cancer as determined by immunohistochemistry (IHC) staining (IHC 1+, 2+, 3+) or next-generation sequencing (NGS) of tissue or circulating tumor DNA (i.e., evaluation of HER2 copy numbers or mutations) (note: documentation of HER2 status is required prior to Screening;
5. In the opinion of the Investigator, is medically confirmed to derive no clinical benefit from other standard therapies.
6. In the opinion of the Investigator, has a life expectancy > 6 months.
7. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 at Screening.
8. Women of childbearing potential (WOCBP) who engage in heterosexual intercourse must agree to maintain effective contraception during the study and for up to 6 months after EOT; males whose sexual partners are WOCBP must also agree to maintain effective contraceptive method and should refrain from donating sperm during the study and for up to 6 months after EOT.

Exclusion Criteria:

1. Has a confirmed HER2 exon 20 mutation (in the documented NGS test result).
2. Received any IP, cytotoxic chemotherapy, or other anticancer drugs from a previous treatment regimen or clinical study within 3 weeks of the first dose of the study IP (note: Rescreening will be permitted after a washout period of 3 weeks).
3. Has been previously treated with systemic anticancer treatment of more than 6 regimens for breast cancer or 3 regimens for other solid tumors (note: local administration of rituximab is allowed but intrathecal methotrexate or concurrent chemoradiotherapy is regarded as systemic therapy).
4. Has any AEs from previous chemotherapy that have not recovered to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Grade ≤ 1 (note: Grade ≤ 2 peripheral neuropathy or hair loss is acceptable).
5. Is a female who is pregnant, breastfeeding, or (among those of childbearing potential) planning to become pregnant.
6. Has a history of other active malignancy within 3 years prior to Screening (note: patients with non-melanoma skin cancer, in situ melanoma, or in situ cervical cancer are permitted to be enrolled).
7. Has any of the following laboratory abnormalities during Screening:

   * Hematology (note: transfusion or hematopoietic growth factor administration within 14 days prior to Screening test is not allowed):

     * -White blood cell (WBC) count < 2.5 × 10 power 9/L
     * -Absolute neutrophil count (ANC) < 1500/µL
     * -Platelets < 100000/µL
     * -Hemoglobin < 9.0 g/dL.
   * Clinical chemistry:

     * -Creatinine clearance < 60 mL/min according to the Cockroft-Gault equation
     * -Total bilirubin > 1.5 × ULN
     * -Aspartate aminotransferase/transaminase (AST or SGOT) > 2.5 × ULN (> 5 × ULN with liver metastases)
     * - Alanine aminotransferase/transaminase (ALT or SGPT) > 2.5 × ULN (> 5 × ULN with liver metastases).
8. Currently has uncontrolled NCI-CTCAE Grade ≥ 2 hypercalcemia.
9. Has undergone prior treatment with a cumulative dose of doxorubicin of > 360 mg/meter square or previous treatment with another anthracycline with a cumulative dose equivalent to > 360 mg/meter square doxorubicin.
10. Has a current infection (including tuberculosis infection, among others) requiring systemic antibacterial, antifungal, or antiviral therapy within 14 days prior to the first dose of the IP (note: antiviral therapy is permitted for patients with hepatocellular carcinoma or chronic hepatitis B virus [HBV] or hepatitis C virus [HCV] infection).
11. Has untreated chronic hepatitis B or is a chronic HBV carrier (undetectable HBV DNA) at Screening (note: patients who are inactive hepatitis B surface antigen [HBsAg] carriers or have treated and stable hepatitis B (undetectable HBV DNA) can be enrolled; patients with detectable HBsAg or detectable HBV DNA should be managed per treatment guidelines. Patients receiving antivirals at Screening should have been treated for > 2 weeks before the first dose of IP).
12. Has active or chronic hepatitis C (note: patients with a negative HCV antibody test at Screening or positive HCV antibody test followed by a negative HCV RNA test at Screening are eligible; the HCV RNA test will only be performed for patients testing positive for HCV antibody. Patients receiving antivirals at Screening should have been treated for > 2 weeks before the first dose of IP).
13. Has a known history of human immunodeficiency virus infection.
14. Has received live vaccines within 4 weeks of the first dose of IP (note: the seasonal flu vaccines that does not contain live virus and coronavirus disease 2019 [COVID-19] vaccines are allowed).
15. Has had major surgery within 4 weeks prior to the first dose of the IP. Patients should have recovered from the effects of major surgery or significant traumatic injury within 16 days prior to the first dose of the IP (note: major surgery is defined as one that cannot be performed with local anesthesia [i.e., general anesthesia, respiratory assistance, or regional anesthesia] or an open biopsy).
16. Has received radiotherapy to a large field or including a vital organ within 14 days prior to the first dose of the IP (or 7 days prior to the first dose of the IP if a vital organ is not included).
17. Has central nervous system (CNS) metastases or spinal cord compression that are associated with progressive neurological symptoms, or that require treatment with more than 10 mg daily of prednisone or equivalent doses of corticosteroids, or that have not been on stable steroid treatment for at least 2 weeks prior to first drug administration (note: CNS metastases that have been either previously treated and controlled, or are symptomatic, or are untreated and asymptomatic are permitted and, when evaluable, should be captured as target lesion).
18. Has any other medical condition (with the exclusion of brain metastases as described above) requiring prednisone therapy of more than 10 mg daily or equivalent systemic steroid therapy (steroid replacement therapy for adrenal or pituitary insufficiency is permitted) or has received treatment with steroids for current or past non-infectious pneumonitis/interstitial lung disease.
19. Has impaired cardiac function or clinically significant cardiac disease, including:

    * New York Heart Association Grade 2 or higher congestive heart failure.
    * Left ventricular ejection fraction < 50% within the last 6 months.
    * Coronary artery bypass graft or vascular stent implantation.
    * Any other uncontrolled cardiac condition such as unstable angina, arrhythmias requiring treatment, atrial fibrillation, or hypertension (systolic blood pressure > 160 mmHg, diastolic blood pressure > 100 mmHg).
    * Baseline prolongation of QT interval corrected for heart rate using Fridericia's method (QTcF) of > 470 msec for females or > 450 msec for males determined (by the average of 3 readings on triplicate 12-lead ECG) or history of long QTc syndrome (congenital or otherwise) or Torsade de Pointes.
20. Is unable to swallow capsules or has intractable nausea, vomiting, or gastrointestinal diseases that interfere with proper absorption, or has any absorption disorders that may interfere with absorption of the IP.
21. Has known or suspected allergy or anaphylaxis to any component of the IP.
22. Has pleural effusion, ascites, or pericardial effusion requiring catheter drainage, peritoneal shunting, or Cell-free and concentrated Ascites Reinfusion Therapy (CART) (note: CART is not allowed within 2 weeks of the Screening visit).
23. Has retinal vascular disorder, retinopathy, glaucoma, or retinal detachment.
24. Any other clinically significant comorbidities, such as neurological or psychological disorders, which in the judgment of the Investigator, could compromise compliance with the protocol, interfere with the interpretation of study results, or predispose the subject to safety risks.
25. For any other reason, as determined by the Investigator, the patient is deemed inappropriate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Estimate of Maximum tolerated dose (MTD) of VRN101099 | Up to 2 years post first dose administration
  This will be based on dose limiting toxicities (DLT) observed during the DLT evaluation period.
Number of participants with Adverse events (AEs) and Serious Adverse events (SAE) as assessed by Medical Dictionary for Regulatory Activities (MedDRA®). | Up to 2 years post first dose administration
Number of patients with changes in ECOG performance status from baseline following treatment with VRN101099 | From Screening to 14 days post last dose
Number of patients with changes in physical/ophthalmic examination from baseline following treatment with VRN101099 | From Screening to 14 days post last dose
Number of patients with changes in laboratory tests from baseline following treatment with VRN101099 | From Screening to 14 days post last dose

SECONDARY OUTCOMES:
Plasma PK of VRN101099 and Cycle1 Day 1- Cmax | Blood sampling from pre dose to 24 hours post dose administration on Cycle1 Day 1 and Day 15 (C1D1, C1D15) and pre dose on Cycle 1 Day 8 (C1D8). Each Cycle-28 days. Additionally, on Predose on Cycle 2 Day 1, Cycle 2 Day 8 and Day 1 of subsequent cycles.
  Cmax- Maximum plasma concentration
Plasma PK of VRN101099 and Cycle1 Day 1-AUC0-last | Blood sampling from pre dose to 24 hours post dose administration on Cycle1 Day 1 and Day 15 (C1D1, C1D15) and pre dose on Cycle 1 Day 8 (C1D8). Each Cycle-28 days. Additionally, on Predose on Cycle 2 Day 1, Cycle 2 Day 8 and Day 1 of subsequent cycles.
  AUC- Area under curve at time 0 to last
Plasma PK of VRN101099 and Cycle1 Day 1-AUC0-Inf | Blood sampling from pre dose to 24 hours post dose administration on Cycle1 Day 1 and Day 15 (C1D1, C1D15) and pre dose on Cycle 1 Day 8 (C1D8). Each Cycle-28 days. Additionally, on Predose on Cycle 2 Day 1, Cycle 2 Day 8 and Day 1 of subsequent cycles.
  AUC- Area under curve at time 0 to Infinity
Plasma PK of VRN101099 and Cycle1 Day 1-Tmax | Blood sampling from pre dose to 24 hours post dose administration on Cycle1 Day 1 and Day 15 (C1D1, C1D15) and pre dose on Cycle 1 Day 8 (C1D8). Each Cycle-28 days. Additionally, on Predose on Cycle 2 Day 1, Cycle 2 Day 8 and Day 1 of subsequent cycles.
  Tmax- Time for maximum concentration
Plasma PK of VRN101099 and Cycle1 Day 1- λz | Blood sampling from pre dose to 24 hours post dose administration on Cycle1 Day 1 and Day 15 (C1D1, C1D15) and pre dose on Cycle 1 Day 8 (C1D8). Each Cycle-28 days. Additionally, on Predose on Cycle 2 Day 1, Cycle 2 Day 8 and Day 1 of subsequent cycles.
  λz- Terminal rate constant
Plasma PK of VRN101099 and Cycle1 Day 1- t1/2 | Blood sampling from pre dose to 24 hours post dose administration on Cycle1 Day 1 and Day 15 (C1D1, C1D15) and pre dose on Cycle 1 Day 8 (C1D8). Each Cycle-28 days. Additionally, on Predose on Cycle 2 Day 1, Cycle 2 Day 8 and Day 1 of subsequent cycles.
  T1/2- Terminal half life
Plasma PK of VRN101099 and Cycle1 Day 1- CL/F | Blood sampling from pre dose to 24 hours post dose administration on Cycle1 Day 1 and Day 15 (C1D1, C1D15) and pre dose on Cycle 1 Day 8 (C1D8). Each Cycle-28 days. Additionally, on Predose on Cycle 2 Day 1, Cycle 2 Day 8 and Day 1 of subsequent cycles.
  CL/F- Apparent plasma clearance
Plasma PK of VRN101099 and Cycle1 Day 15- Cmax,ss | Blood sampling from pre dose to 24 hours post dose administration on Cycle1 Day 1 and Day 15 (C1D1, C1D15) and pre dose on Cycle 1 Day 8 (C1D8). Each Cycle-28 days. Additionally, on Predose on Cycle 2 Day 1, Cycle 2 Day 8 and Day 1 of subsequent cycles.
  Cmax, ss- Maximum plasma concentration at steady state
Plasma PK of VRN101099 and Cycle1 Day 15- Cmin,ss | Blood sampling from pre dose to 24 hours post dose administration on Cycle1 Day 1 and Day 15 (C1D1, C1D15) and pre dose on Cycle 1 Day 8 (C1D8). Each Cycle-28 days. Additionally, on Predose on Cycle 2 Day 1, Cycle 2 Day 8 and Day 1 of subsequent cycles.
  Cmin, ss- Minimum drug concentration at steady-state
Plasma PK of VRN101099 and Cycle1 Day 15- Tmax,ss | Blood sampling from pre dose to 24 hours post dose administration on Cycle1 Day 1 and Day 15 (C1D1, C1D15) and pre dose on Cycle 1 Day 8 (C1D8). Each Cycle-28 days. Additionally, on Predose on Cycle 2 Day 1, Cycle 2 Day 8 and Day 1 of subsequent cycles.
  Tmax,ss Time for maximum concentration at steady-state
Plasma PK of VRN101099 and Cycle1 Day 15- AUC 0-last | Blood sampling from pre dose to 24 hours post dose administration on Cycle1 Day 1 and Day 15 (C1D1, C1D15) and pre dose on Cycle 1 Day 8 (C1D8). Each Cycle-28 days. Additionally, on Predose on Cycle 2 Day 1, Cycle 2 Day 8 and Day 1 of subsequent cycles.
  AUC 0-last- Area under curve 0 to last
Plasma PK of VRN101099 and Cycle1 Day 15- swing | Blood sampling from pre dose to 24 hours post dose administration on Cycle1 Day 1 and Day 15 (C1D1, C1D15) and pre dose on Cycle 1 Day 8 (C1D8). Each Cycle-28 days. Additionally, on Predose on Cycle 2 Day 1, Cycle 2 Day 8 and Day 1 of subsequent cycles.
Plasma PK of VRN101099 and Cycle1 Day 15- Fluctuation | Blood sampling from pre dose to 24 hours post dose administration on Cycle1 Day 1 and Day 15 (C1D1, C1D15) and pre dose on Cycle 1 Day 8 (C1D8). Each Cycle-28 days. Additionally, on Predose on Cycle 2 Day 1, Cycle 2 Day 8 and Day 1 of subsequent cycles.
Plasma PK of VRN101099 and Cycle1 Day 15- Ctrough | Blood sampling from pre dose to 24 hours post dose administration on Cycle1 Day 1 and Day 15 (C1D1, C1D15) and pre dose on Cycle 1 Day 8 (C1D8). Each Cycle-28 days. Additionally, on Predose on Cycle 2 Day 1, Cycle 2 Day 8 and Day 1 of subsequent cycles.
To evaluate objective response rate (ORR) | Up to 2 years post first dose administration
  The proportion of patients whose best overall response (BOR) is either confirmed complete responses (CR) or confirmed partial responses (PR).
Number of patients with disease Control Rate (DCR) | Up to 2 years post first dose administration
  Percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease to a therapeutic intervention in clinical trials of anticancer agents.
Number of patients with changes in duration of objective response (DOR) | Up to 2 years post first dose administration
  The time from first documented disease control response (confirmed CR, confirmed PR, or confirmed SD) until the earlier of disease progression or death from any cause, whichever occurs first. This will only be applicable for patients who have a confirmed best overall response of CR, PR, or SD. Patients without the events (progressive disease or death) will be censored at the date of their last tumor assessment
To assess progression-free survival (PFS) | Up to 2 years post first dose administration
  The time from start of study treatment to the earlier of either disease progression or death from any cause, whichever occurs first.
To assess time to progression (TTP) | Up to 2 years post first dose administration
  TTP- Time between the starting time and local tumor progression per tumor treated.

CONTACTS AND LOCATIONS:
Overall Officials: Daekwon Kim, Study Chair — Voronoi, Inc. Chief Executive Officer
Locations (1):
- St Vincent's Hospital Sydney, Darlinghurst, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No